CLINICAL TRIAL: NCT01853943
Title: Hand Grip Test After Transradial Percutaneous Coronary Procedures
Brief Title: Hand Grip Test and Transradial Coronary Procedures
Acronym: HANGAR
Status: Completed | Type: Observational
Sponsor: Ospedale Sandro Pertini, Roma (Other)
Responsible Party: Principal Investigator, Alessandro Sciahbasi, MD, MD, Ospedale Sandro Pertini, Roma
Other Study IDs: Pertini-02
Record Dates: First submitted 2013-05-10; First posted 2013-05-15 (Estimated); Last update posted 2015-03-03 (Estimated); Status verified 2015-03

CONDITIONS: Radial Artery Occlusion
Keywords: Transradial approach; radial occlusion; hand grip; coronary angiography
MeSH Terms: conditions — Arterial Occlusive Diseases; Bites and Stings

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patent radial artery: Patient with patent radial artery after the percutaneous coronary procedure
- Occluded radial artery: Patients with occluded radial artery after the procedure

SUMMARY:
Transradial coronary procedures are gaining in popularity worldwide. A possible complication of transradial approach is the occlusion of the radial artery that in most cases is asymptomatic. However the investigators do not know if the radial artery occlusion may impact over the muscle force of the hand or fingers.

To evaluate if transradial approach for percutaneous coronary procedures may affect muscle force of the hand, thumb and index finger the investigators use a standardized hand-grip manometer and a pinch gauge before the transradial procedure, the day after the procedures and after few months.

ELIGIBILITY:
Inclusion Criteria:

Stable patients who undergo elective percutaneous transradial coronary procedures

Exclusion Criteria:

* hemodynamic instability,
* acute coronary syndromes,
* haemodialysis patients with an arteriovenous fistula,
* sheath diameter > 6 French,
* age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stable patients who undergo elective percutaneous transradial coronary procedures
Sampling Method: Non-Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2012-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Hand grip strength | 3 months
  The variation in had grip strength and thumb pinch after the procedure (the day after and at 30 day follow-up) compared to baseline in patients with patent radial artery compared to occluded radial artery.

SECONDARY OUTCOMES:
Radial occlusion | 3 months
  The rate of radial occlusion after transradial coronary procedures

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Sciahbasi, MD, Principal Investigator — Ospedale Sandro Pertini - ASL RMB
Locations (1):
- Ospedale Sandro Pertini - ASL RMB, Rome, Italy